CLINICAL TRIAL: NCT07142993
Title: Impact of Social Media-Based Networked Follow-up Nursing Intervention on Itch Severity and Self-care Ability in Patients With Atopic Dermatitis
Brief Title: Social Media Follow-up Nursing for Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Ruimin Wang, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-S-0038
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Social Media-Based Nursing Intervention Group (Experimental): Patients (n=50) received networked follow-up nursing intervention via a popular social media platform (WeChat). This included weekly educational materials, daily Q&A sessions, personalized care plans, remote monitoring of skin condition via photos, continuous health education, and a peer communication group. This intervention was provided as an adjunct to standard medical care.
  Interventions: Behavioral: Social Media-Based Nursing Intervention
- Active Comparator: Conventional Nursing Care Group (Active Comparator): Patients (n=50) received conventional nursing care. This included verbal health education at discharge, distribution of educational materials and a follow-up handbook, and weekly follow-up phone calls from a liaison nurse to assess adherence and provide guidance. This intervention was provided as an adjunct to standard medical care.
  Interventions: Behavioral: Conventional Nursing Care

INTERVENTIONS:
Behavioral: Social Media-Based Nursing Intervention — A structured nursing follow-up program delivered through a WeChat group. The program included regular sharing of educational content (articles, videos), personalized care advice, remote photo-based monitoring by medical staff, and peer support within the group. The intervention was managed by a dedicated team of dermatologists and nurses.
  Arms: Experimental: Social Media-Based Nursing Intervention Group
Behavioral: Conventional Nursing Care — A standard care follow-up protocol involving verbal education at discharge, provision of printed health materials, and proactive weekly telephone calls to monitor the patient's condition, correct improper self-care actions, and encourage clinic visits if necessary.
  Arms: Active Comparator: Conventional Nursing Care Group

SUMMARY:
This is a randomized controlled study to evaluate the effectiveness of a social media-based (WeChat) networked nursing follow-up intervention compared to conventional nursing care for patients with atopic dermatitis. The study aims to determine the impact of the intervention on itch severity, skin condition, and self-care ability over a 6-month period.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic, relapsing inflammatory skin disease that requires long-term management. Traditional outpatient care is often insufficient for managing the chronic nature of the disease. This study explores the effects of social media-based networked follow-up nursing interventions, leveraging popular platforms like WeChat to provide continuous support, personalized care plans, remote monitoring, and health education. This study prospectively enrolled and randomized 100 patients with AD into two groups: a research group receiving the social media-based intervention and a control group receiving conventional nursing care. The primary objective is to compare the differences in itch severity, eczema area and severity index (EASI), overall disease assessment (IGA), and self-care ability between the two groups from baseline to 6 months post-intervention. The study aims to provide evidence for social media-based nursing as an effective adjunctive management strategy for improving outcomes in patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-60 years;
2. Diagnosed according to the Williams diagnostic criteria for atopic dermatitis;
3. Signed informed consent.

Exclusion Criteria:

1. Severe, progressive, and uncontrolled major organ or systemic diseases (including cardiovascular, liver, lung, and kidney diseases), other autoimmune diseases, or malignant tumors;
2. Pregnant or lactating women;
3. Presence of other skin diseases;
4. Mental health disorders;
5. Previous experience with similar follow-up nursing interventions;
6. Severe complications such as infections or allergies.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Itch Severity | Baseline, 6 Months
  Measured by the Numeric Rating Scale (NRS) for itching. The scale ranges from 0 (no itching) to 10 (very severe itching), where patients rate the most severe itching experienced in the past 24 hours. A higher score indicates more severe itching.
Change in Self-care Ability | Baseline, 6 Months
  Measured by the Exercise of Self-Care Agency Scale (ESCA). The scale includes 43 items across four dimensions (self-care skills, self-responsibility, self-concept, and health knowledge). It uses a Likert 5-point scoring system (0 to 4 points). A higher total score indicates stronger self-care ability.

SECONDARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | Baseline, 6 Months
  EASI is used to evaluate the eczema area and severity. It assesses four clinical signs (erythema, papules/edema, lichenification, epidermal peeling) on a scale of 0 to 3 based on severity. A higher score indicates greater disease severity.
Change in Overall Evaluation Score | Baseline, 6 Months
  Measured by the Investigator's Global Assessment (IGA). A six-level scoring system (0 to 5) is used, where 0 indicates no lesions and 5 indicates very severe disease. A higher score indicates greater overall disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China